CLINICAL TRIAL: NCT01157663
Title: The Effect of Balance Training in People With Functional Ankle Instability
Brief Title: The Effect of Balance Training in People With Functional Ankle Instability (FAI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/345
Record Dates: First submitted 2010-06-30; First posted 2010-07-07 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Functional Ankle Instability
Keywords: Functional ankle instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adapted Balance Training group (Experimental)
  Interventions: Other: Adapted balance training
- Standard Balance training group (Active Comparator): Balance training with unipedal standing during 8 weeks
  Interventions: Other: Balance Training

INTERVENTIONS:
Other: Adapted balance training — during 8 weeks
  Arms: Adapted Balance Training group
Other: Balance Training — Balance training with unipedal standing during 8 weeks
  Arms: Standard Balance training group

SUMMARY:
Ankle sprain is the most occurring sport related injury. In addition, 40% of the people who sustain such an injury display residual symptoms under the general denominator functional ankle instability (FAI). In literature, there is already given a lot of attention to extrinsic and intrinsic risk factors of FAI. Furthermore, there is a major focus on the possible interventions which may be able to reduce the chance of developing chronic instability. At this moment there is a lack of unequivocality.

In this study the investigators address the question of what is the effect of a balance training programme on the movement strategy. Therefore kinematics, kinetics, plantar pressure measurements and muscle activity are taken in consideration The purpose of this study is a better insight in the effect of treatment on the residual symptoms related to FAI.

ELIGIBILITY:
Inclusion Criteria:

* a history of more than 1 unilateral ankle sprain
* presence of feeling of 'giving way'
* a feeling of weakness around the ankle
* a decreased functional participation

Exclusion Criteria:

* ankle fracture
* ankle surgery
* lower limb pain (not related to an ankle sprain)
* ankle distortion in the last 3 months
* currently receiving treatment
* disturbance of equilibrium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
effect of balance training on movement strategy | after 8 weeks of treatment
  kinematics, kinetics, plantar pressures and muscle activity

SECONDARY OUTCOMES:
self-assessed complaints registration using questionnaires | after 8 weeks
self-assessed complaints registration using questionnaires | after 1 year
self-assessed complaints registration using questionnaires | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Philip Roosen, PhD, Principal Investigator — University Ghent
Locations (1):
- University Ghent, Ghent, Belgium